CLINICAL TRIAL: NCT05475015
Title: Three-dimensional MR Elastography for Assessing Cirrhosis and Portal Hypertension (CHESS2206): A Prospective Multicenter Study
Brief Title: 3D-MRE for Assessing Cirrhosis, Advanced Chronic Liver Disease and Portal Hypertension
Status: Recruiting | Type: Observational
Sponsor: Shengjing Hospital (Other)
Collaborators: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Yu Shi, Deputy director of department of radology, Shengjing Hospital
Other Study IDs: CHESS2206
Record Dates: First submitted 2022-07-19; First posted 2022-07-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-12

CONDITIONS: Cirrhosis, Liver; Portal Hypertension; Advanced Chronic Liver Disease
Keywords: 3D-MRE; HVPG; advanced chronic liver disease
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort: Training cohort was set to develop the novel non-invasive model for virtual HVPG
  Interventions: Device: 3D-MRE; Device: HVPG
- Validation cohort: Validation cohort was set to validate the novel non-invasive model for virtual HVPG in different people in same environments
  Interventions: Device: 3D-MRE; Device: HVPG

INTERVENTIONS:
Device: 3D-MRE — All imaging studies were performed by using a 3.0-T MRI system ( GE Healthcare) with a phasedarray body coil.
Device: HVPG — HVPG measurements are performed by well-trained interventional radiologists in accordance with standard operating procedures.

SUMMARY:
How to construct a novel, non-invasive, accurate, and convenient method to achieve prediction of hepatic venous pressure gradient (HVPG) is an important general problem in the management of portal hypertension in cirrhosis or advanced chronic liver disease. We plan to investigate the ability of three demensional-magnetic resonance elastography (3D-MRE) to establish a risk stratification system and perform tailored management for portal hypertension in cirrhosis or advanced chronic liver disease.

DETAILED DESCRIPTION:
China suffers the heaviest burden of liver disease in the world. The number of chronic liver disease is more than 400 million. Either viral-related hepatitis, alcoholic hepatitis, or metabolic-related fatty hepatitis, etc. may progress to cirrhosis, which greatly threatens public health. Portal hypertension is a critical risk factor that correlates with clinical prognosis of patients with cirrhosis. According to the Consensus on clinical application of hepatic venous pressure gradient in China (2018), hepatic venous pressure gradient (HVPG) greater than 10,12,16,20 mmHg correspondingly predicts different outcomes of patients with cirrhosis portal hypertension. It is of great significance to establish a risk stratification system and perform tailored management for portal hypertension in cirrhosis. As a universal gold standard for diagnosing and monitoring portal hypertension, HVPG remains limitation for clinical application due to its invasiveness. How to construct a novel, non-invasive, accurate, and convenient method to achieve prediction of HVPG is an important general problem in the management of portal hypertension in cirrhosis and advanced chronic liver disease.

Multiparametric three-dimensional (3D) MR elastography allows for basic viscoelastic modeling of tissue, partitioning the complex shear modulus into elastic components (eg, storage modulus) and viscous components (eg, loss modulus and damping ratio [DR]). However, these mechanical properties of tissue measured with use of 3D MR elastography have yet to be investigated in cirrhosis to identify specific hepatic pathophysiologic interrelations. We hypothesize that these mechanical properties might be valid presumptive surrogates of cirrhosis and portal hypertension, perhaps capable of supplanting liver biopsy or other invasive diagnostic interventions. This project aims to investigate the ability of three demensional-magnetic resonance elastography (3D-MRE) to establish a risk stratification system and perform tailored management for portal hypertension in cirrhosis and advanced chronic liver disease.

ELIGIBILITY:
Inclusion criteria were: (1) ≥18 years; (2) written informed consent; (3) confirmed ACLD of any liver disease etiology; (4) clinically indicated for HVPG measurement, with 3D-MRE performed within one month prior.

Exclusion criteria were: (1) hepatic or extrahepatic malignancies, or large hepatic or splenic focal diseases affecting MRE measurement; (2) MR or HVPG contraindications; (3) prior liver or splenic surgery affecting MRE measurement; (4) treatment with nonselective β-blockers (NSBB) between MRE and HVPG measurements; (5) invalid or unreliable HVPG or MRE results and (6) biliary obstruction or dilation on MR images.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Organize paticipating units to collect standard-of-care data including radiological and clinical data. Patients diagnosed with cirrhosis who received HVPG measurement and 3D-MRE should be enrolled.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the features of 3D-MRE for assessing portal hypertension in cirrhosis. | 12 months
  WIth HVPG as reference standand, the overall diagnostic perforemace (accuracy) for cirrhosis and portal hypertension of 3D-MRE was assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Shi, Prof., Principal Investigator — Shengjing Hospital; Shenghong Ju, Prof., Principal Investigator — Zhongda Hospital; Xiaolong Qi, Prof., Principal Investigator — Zhongda Hospital
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shi Y, Qi YF, Lan GY, Wu Q, Ma B, Zhang XY, Ji RY, Ma YJ, Hong Y. Three-dimensional MR Elastography Depicts Liver Inflammation, Fibrosis, and Portal Hypertension in Chronic Hepatitis B or C. Radiology. 2021 Oct;301(1):154-162. doi: 10.1148/radiol.2021202804. Epub 2021 Aug 10. PMID 34374594
- [Background] Yu Q, Huang Y, Li X, Pavlides M, Liu D, Luo H, Ding H, An W, Liu F, Zuo C, Lu C, Tang T, Wang Y, Huang S, Liu C, Zheng T, Kang N, Liu C, Wang J, Akcalar S, Celebioglu E, Ustuner E, Bilgic S, Fang Q, Fu CC, Zhang R, Wang C, Wei J, Tian J, Ormeci N, Ellik Z, Asiller OO, Ju S, Qi X. An imaging-based artificial intelligence model for non-invasive grading of hepatic venous pressure gradient in cirrhotic portal hypertension. Cell Rep Med. 2022 Mar 15;3(3):100563. doi: 10.1016/j.xcrm.2022.100563. eCollection 2022 Mar 15. PMID 35492878